CLINICAL TRIAL: NCT06086704
Title: Phase II Study of 18F-FFNP Breast PET/MRI in the Assessment of Early Response of Breast Cancer to Presurgical Endocrine Therapy
Brief Title: Study of 18F-FFNP Breast PET/MRI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-1114; Protocol Version 7/30/2024 (Other: UW Madison); SMPH/RADIOLOGY/RADIOLOGY (Other: UW Madison); UW23020 (Other: UWCCC OnCore ID); 1R01CA272571-01 (NIH)
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: PR+
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging; Anastrozole; Blood Specimen Collection; gadopiclenol

STUDY DESIGN:
Intervention Model Description: Window of Opportunity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Metabolite Analysis (Experimental): participants will undergo venous blood sampling during the PET/MRI scan
  Interventions: Drug: 18F-fluorofuranylnorprogesterone; Device: Positron Emissions Tomography / Magnetic Resonance Imaging; Other: Blood Sampling; Drug: FDA-approved gadolinium-based intravenous contrast agent
- Group 2: Pre-surgical Treatment (Experimental): participants will undergo PET/MRI scans before and after 2 weeks treatment with anastrozole
  Interventions: Drug: 18F-fluorofuranylnorprogesterone; Device: Positron Emissions Tomography / Magnetic Resonance Imaging; Drug: Anastrozole; Drug: FDA-approved gadolinium-based intravenous contrast agent
- Group 3: Test-Retest (Experimental): participants will undergo baseline and repeat PET/MRI scans without intervening treatment to determine repeatability
  Interventions: Drug: 18F-fluorofuranylnorprogesterone; Device: Positron Emissions Tomography / Magnetic Resonance Imaging; Drug: FDA-approved gadolinium-based intravenous contrast agent

INTERVENTIONS:
Drug: 18F-fluorofuranylnorprogesterone — 18F-FFNP will be given by a slow infusion (approximately 2 minutes), and the dose administered will be approximately 7 mCi.
  Other Names: FFNP
Device: Positron Emissions Tomography / Magnetic Resonance Imaging — Breast specific PET/MRI data will be acquired using a 3T simultaneous PET/MRI scanner (Signa PET/MR, GE Healthcare)
  Other Names: PET/MRI
Drug: Anastrozole — hormone based chemotherapy that reduces estrogen, 1 mg anastrozole once daily by mouth for a minimum of 14 days
  Arms: Group 2: Pre-surgical Treatment
Other: Blood Sampling — Venous blood samples will be collected at multiple timepoints (e.g., 5, 10, 20, 30, and 45 min after 18F-FFNP injection to determine parent and metabolite fractions
  Arms: Group 1: Metabolite Analysis
Drug: FDA-approved gadolinium-based intravenous contrast agent — FDA-approved gadolinium-based intravenous contrast agent used for the MRI portion of this study
  Other Names: gadopiclenol; gadobenate dimuglumine

SUMMARY:
This clinical trial will investigate an estrogen-regulated parameter as an early measure of endocrine therapy response: progesterone receptor (PR) protein with a progestin-based radioligand, 18F-fluorofuranylnorprogesterone (18F-FFNP). The overall purpose of this research is to test the efficacy of 18F-FFNP PET/MRI for predicting response to presurgical endocrine therapy and to determine the quantitative reliability of 18F-FFNP breast PET/MRI in patients with newly diagnosed PR+ primary breast cancer.

DETAILED DESCRIPTION:
Primary Objective

• Determine the diagnostic accuracy of 18F-FFNP PET/MRI for predicting response to presurgical endocrine therapy.

Secondary Objectives

* Determine the repeatability of quantitative assessment of tumor 18F-FFNP uptake.
* Determine the intra- and inter-observer variability of quantitative assessment of tumor 18F-FFNP uptake.
* Assess the safety and tolerability of 18F-FFNP.

Exploratory Objectives

* Define the parent and metabolite fractions of 18F-FFNP over the time course of the scan.
* Assess the association between tumor 18F-FFNP uptake with serum progesterone, estradiol, and corticosteroid binding globulin levels.
* Compare changes in 18F-FFNP breast PET/MRI parameters with changes in PR immunohistochemistry in therapy responders and non-responders.
* Assess the association between tumor 18F-FFNP uptake with disease recurrence.
* Determine whether MRI parameters improve the predictive value of FFNP PET alone.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal status defined by either

  * prior bilateral oophorectomy
  * age greater than or equal to 60 years of age
  * age less than 60 years of age and amenorrheic for 12 or more months in the absence of prior chemotherapy, tamoxifen, toremifene or ovarian suppression and FSH and estradiol in the postmenopausal range per local normal range (Group 2 only)
* Diagnosis of biopsy-proven invasive breast cancer measuring at least 1.0 cm in diameter by any imaging modality
* Biopsy-proven PR-positive invasive breast cancer
* Breast MRI planned or performed before surgery
* Definitive surgical excision of the primary tumor planned without neoadjuvant therapy; defined as therapy (chemotherapy, targeted therapy, radiation therapy or endocrine therapy) given to decrease the size of the tumor prior to planned surgery.

Exclusion Criteria:

* Inability or unwillingness to provide informed consent to the study
* HER2-positive breast cancer, as defined by immunohistochemical staining 3+ OR positive by in situ hybridization (Group 2 only)
* PR and Ki67 IHC slides or FFPE tissue blocks from clinical breast biopsy not available
* Patients who have completed neoadjuvant chemotherapy, endocrine therapy, targeted therapy, surgical resection, or radiation for the current biopsy-proven malignancy
* Patients who are planning to undergo anastrozole as standard of care neoadjuvant therapy
* Patients who are currently taking aromatase inhibitors or ER antagonists (tamoxifen, raloxifene)
* Patients with breast expanders
* Patients who are pregnant or lactating
* Patients with a contraindication to gadolinium-based contrast agents, including allergy or impaired renal function (per UW Health Guidelines)
* Patients with a history of allergic reaction attributable to compounds of similar chemical or biologic composition to 18F-FFNP
* Patients with history of allergic reaction to anastrozole (Group 2 only)
* Patients in liver failure as judged by the patient's physician
* Patients with standard contraindications to MRI (per UW Health Guidelines)
* Patients requiring conscious sedation for imaging are not eligible; patients requiring mild, oral anxiolytics for the clinical MRI scan will be allowed to participate as long as the following criteria are met:

  * The patient has their own prescription for the medication
  * The informed consent process is conducted prior to the self-administration of the medication.
  * The patient comes to the research visit with a driver.
* Patients unable to lie prone for 45 minutes for imaging
* Patients taking hormone replacement therapy or over-the-counter products/supplements/herbal preparation with potential estrogenic effects who are unwilling to discontinue these agents during the timeframe of the study until surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Percentage change in 18F-FFNP uptake between baseline and follow-up PET/MRI scans | up to 4 weeks on study and up to 7 weeks on study
  Tumor uptake values of 18F-FFNP will be obtained from the attenuation corrected PET component of the simultaneous breast 18F-FFNP PET/MRI research scan according to the procedures detailed in the imaging manual and the FDA IND.
Percentage change in tumor Ki67 proliferation score, as a surrogate measure of endocrine sensitivity | up to 4 weeks on study and up to 7 weeks on study
  Baseline Ki67 proliferation immunohistochemistry score will be obtained from the existing clinical standard-of-care breast biopsy. Post-treatment K67 proliferation immunohistochemistry score will be obtained from the surgical specimen after excision.
  Treatment response is defined as a reduction in Ki67 score of greater than or equal to 60 percent. Treatment nonresponse is defined as a reduction of less than 60 percent.

SECONDARY OUTCOMES:
Qualitative Analysis of 18F-FFNP uptake | imaging takes up to 2 hours during a visit and will take place up to 4 weeks and up to 6 weeks for the test-retest Group 3
  18F-FFNP uptake will be visually evaluated qualitatively with the following grading scale: no uptake (tumor < background), minimal uptake (tumor = background), mild (tumor slightly > background), moderate uptake (tumor >> background), and intense uptake (tumor >>> background). Tumor uptake will also be dichotomized as increased (mild, moderate, or intense uptake) or absent (no uptake, minimal).
Intra- and Inter-Observer Variability of Quantitative Assessment of Tumor 18F-FFNP uptake | imaging takes up to 2 hours during a visit and will take place up to 4 weeks and up to 6 weeks for the test-retest Group 3
  For the test-retest portion of the clinical trial, the mixed effects model framework will be utilized to determine the intra- and interobserver variability of quantitative assessment of tumor 18F-FFNP uptake via a parametric bootstrapping approach.
Quantitative Assessment of Tumor 18F-FFNP: Standardized Uptake Values (SUV) | imaging takes up to 2 hours during a visit and will take place up to 4 weeks and up to 6 weeks for the test-retest Group 3
  Differences in repeatability of the different SUV measures (SUVmax, SUVpeak, and SUVmean) and their respective methods of normalization will be assessed by comparing the variances of the relative test-retest differences, using the Pitnam-Morgan test for correlated variances.
Test-Retest Variability of Quantitative Assessment of Tumor 18F-FFNP uptake | imaging takes up to 2 hours during a visit and will take place up to 4 weeks and up to 6 weeks for the test-retest Group 3
  For the test-retest portion of the clinical trial, the mixed effects model framework will be utilized to determine the test-retest variability of quantitative assessment of tumor 18F-FFNP uptake via a parametric bootstrapping approach.
NCIC Adverse Events Version 5.0 Frequency Tables | up to 7 weeks
  Safety and tolerability of 18F-FFNP by NCIC Adverse Events Version 5.0 will be assessed by frequency tables and possible relationship to study drug as assessed by the investigators.

OTHER OUTCOMES:
Summary of Parent and Metabolite Fractions of 18F-FFNP over the course of the scan | imaging takes up to 2 hours during a visit and will take place up to 4 weeks on study for Group 1
  Median and interquartile ranges will be calculated for metabolized and unmetabolized (parent) 18F-FFNP obtained from subjects undergoing venous blood sampling in the metabolite study and plotted against time.
Statistical Correlation between tumor 18F-FFNP uptake with serum progesterone, estradiol, and corticosteroid binding globulin levels | imaging takes up to 2 hours during a visit and will take place up to 4 weeks on study for Group 1
  Pearson's or Rank correlation analysis will be performed to assess the association between tumor 18F-FFNP uptake with serum progesterone, estradiol, and corticosteroid binding globulin levels. Scatter plots, correlation coefficients (rho), 95% confidence intervals, and p values will be reported.
Statistical correlation between 18F-FFNP breast PET/MRI parameters and changes in PR immunohistochemistry in therapy responders and non-responders | imaging takes up to 2 hours during a visit and will take place up to 4 weeks on study for Group 1, up to 4 weeks and up to 7 weeks for Group 2, and up to 4 weeks and up to 6 weeks for Group 3
  An ANCOVA model, which will include treatment as a fixed effect and the corresponding baseline value as a covariate, and a paired t-test will be utilized to compare the change in tumor 18F-FFNP update after window treatment with change in PR immunostaining from the biopsy to surgical specimen. Means and standard errors will be presented. Least-squares means and 95% CI will be reported. Furthermore, correlation analyses will be performed to describe these associations.
Statistical correlation between tumor 18F-FFNP uptake with disease recurrence | up to 5 years (long term follow up)
  If there is sufficient follow-up data for disease recurrence, the Kaplan-Meier method will be used to analyze time to disease recurrence, defined as date of imaging day until disease recurrence. Patients who do not experience disease recurrence will be censored at the date of last available follow-up. A Cox proportional hazards model will be used to evaluate the association of tumor 18F-FFNP uptake with time to disease recurrence. If there is insufficient follow-up data, descriptive statistics will be used to summarize tumor 18F-FFNP uptake for those patients with disease recurrence
Statistical determination of whether MRI parameters improve the predictive value of FFNP PET alone | up to 5 years (long term follow up)
  The investigators will explore whether adding MRI parameters improves the AUC of 18F-FFNP PET alone. Regression models will be performed on the following parameters: quantitative tumor perfusion (signal enhancement ratio, functional tumor volume), quantitative tumor diffusion (apparent diffusion coefficient), qualitative morphologic phenotype (categories I, II, III, IV), and qualitative background parenchymal enhancement (categories are minimal, mild, moderate, marked).

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Fowler, MD, PHD, Principal Investigator — UW Carbone Cancer Center
Locations (1):
- UW Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No